CLINICAL TRIAL: NCT02224807
Title: Exploring Effects of Weight Loss on Ductal Carcinoma In Situ
Brief Title: Effects of Diet and Exercise on Ductal Carcinoma in Situ
Acronym: DCIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Wendy Demark-Wahnefried, PhD, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: R21CA178359-01A1 (NIH)
Record Dates: First submitted 2014-08-19; First posted 2014-08-25 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Ductal Carcinoma In Situ; Breast Cancer
Keywords: breast cancer; diet; exercise; weight loss
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Breast Neoplasms; Motor Activity; Weight Loss | interventions — Hypoxanthine Phosphoribosyltransferase; Diet; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Progressive Resistance Training (PRT) and a healthy diet (Active Comparator): PRT will be done with resistance bands; participants will receive instruction on three resistance band exercises (triceps, biceps, and shoulder overhead) from an American College of Sports Medicine (ACSM) certified exercise specialist. Participants also will receive dietary counseling from a registered dietitian on correcting nutrient deficiencies that are detected during analysis of their 2-day dietary recalls.
  Interventions: Behavioral: Active Comparator: Progressive Resistance Training (PRT) and a healthy diet
- PRT and a healthy diet, plus weight loss (Experimental): This arm will receive all components of the active comparator arm, plus counseling to achieve a weight loss of 1.5-2 pounds/week. Participants will be trained on how to achieve this caloric deficit through both dietary restriction and increased physical activity. Weight loss will be promoted via a healthy, nutritionally adequate diet consistent with American Cancer Society guidelines. Protein levels will be based on 0.8 g/kg body weight. The distribution of food groups will be customized for preferences. An exercise program will be tailored taking into account kcal expenditure for various activities at a specific body weight; expenditures of 200-400 kcal/day will serve as a goal. Aerobic training of large muscles (legs) will be emphasized to achieve a greater kcal deficit; ramping of intensity and volume over time will be pursued as per the ACSM guidelines. Participants will train once weekly while supervised by an exercise physiologist and daily at home.
  Interventions: Behavioral: Experimental: PRT and a healthy diet, plus weight loss

INTERVENTIONS:
Behavioral: Active Comparator: Progressive Resistance Training (PRT) and a healthy diet — no additional information; see arm description
  Other Names: Diet; Exercise; Physical activity
  Arms: Progressive Resistance Training (PRT) and a healthy diet
Behavioral: Experimental: PRT and a healthy diet, plus weight loss — no additional information, see arm description
  Other Names: Diet; Exercise, Physical Activity
  Arms: PRT and a healthy diet, plus weight loss

SUMMARY:
This pilot/feasibility trial seeks to explore whether an acute bout of negative energy balance prior to surgery affects biomarkers of neoplasia. Forty overweight or obese postmenopausal women diagnosed with ductal carcinoma in situ (DCIS) or early stage breast cancer (Stage I or II) who elect mastectomy or lumpectomy will be randomly assigned to 1-of-2 study arms: 1) an Attention Control Group that receives instruction on dietary approaches to correct nutritional deficiencies and progressive resistance training (PRT) that targets the arm ipsilateral to the affected breast; or 2) an Experimental Group that will receive PRT and guidance to correct nutritional deficiencies plus an intensive intervention to promote a 1.5-2 pound/week weight loss through diet, exercise, and behavior modification. This study will explore and contrast changes in body mass index (BMI) observed from enrollment to the time of surgery in the experimental vs. attention control arms, and also monitor changes in energy intake and physical activity. These changes will be studied in relation to the following endpoints: a) changes in select circulating biomarkers and gene expression related to cancer progression, hormonal status, inflammation and other energy-related factors; b) rates of tumor proliferation and apoptosis; c) tumor markers, e.g., insulin receptor, Vascular Epithelial Growth Factor (VEGF), Nuclear Factor kappa beta (NFkB), and phosphoproteins associated with the Convergence of Hormones, Inflammation and Energy-Rated Factors (CHIEF) pathway; and d) functional and health-related outcomes. Because both tumor tissue and blood will be examined from pre-to-post-intervention, this study will provide exciting new data that can elucidate pathways by which energy balance affects breast cancer progression. Although longer term weight loss is recommended for overweight and obese breast cancer survivors, it is not known whether placing the body in a state of negative energy balance will have a favorable impact on the tumor. If beneficial changes in tumor biology and the host environment occur with short-term, pre-surgical weight loss, this study provides proof of concept that weight loss may offer an acceptable and complementary treatment option that could be combined with standard therapies.

DETAILED DESCRIPTION:
Obesity is a known risk factor for invasive breast cancers that occur post-menopause. Obese women also die twice as frequently from breast cancer than those of normal weight. Numerous preclinical studies show the benefits of caloric restriction on cancer progression in animals - but, will similar effects be seen in humans? In response to a call for translational studies that will identify biological/biobehavioral pathways through which weight loss may affect cancer prognosis (PAR-12-229), the investigators propose a pilot study that builds on the investigators success of pre-surgical interventions to answer the research question, "does negative energy balance with concomitant weight loss invoke anti-cancer effects on tumor biology and the host environment?" The investigators will randomly assign 40 overweight or obese postmenopausal women diagnosed with ductal carcinoma in situ (DCIS) or early stage breast cancer who elect mastectomy or lumpectomy to 1-of-2 study arms: 1) an Attention Control Group that receives instruction on dietary approaches to correct nutritional deficiencies and progressive resistance training (PRT) that targets the arm ipsilateral to the affected breast; or 2) an Experimental Group that will receive PRT and guidance to correct nutritional deficiencies plus an intensive intervention to promote a 1.5-2 pound/week weight loss through diet, exercise, and behavior modification. This study will explore and contrast changes in body mass index (BMI) observed from enrollment to the time of surgery in the experimental vs. attention control arms, and also monitor changes in energy intake and physical activity. These changes will be studied in relation to the following endpoints: a) changes in select circulating biomarkers and gene expression related to cancer progression, hormonal status, inflammation and other energy-related factors; b) rates of tumor proliferation and apoptosis; c) tumor markers, e.g., insulin receptor, Vascular Epithelial Growth Factor (VEGF), Nuclear Factor kappa beta (NFkB), and phosphoproteins associated with the Convergence of Hormones, Inflammation and Energy-Rated Factors (CHIEF) pathway; and d) functional and health-related outcomes. Because both tumor tissue and blood will be examined from pre-to-post-intervention, this study will provide exciting new data that can elucidate pathways by which energy balance affects breast cancer progression from a non-invasive to an invasive state. Although longer term weight loss is recommended for overweight and obese breast cancer survivors, it is not known whether placing the body in a state of negative energy balance will have a favorable impact on the tumor. If beneficial changes in tumor biology and the host environment occur with short-term, pre-surgical weight loss, this study provides proof of concept that weight loss may offer an acceptable and complementary treatment option that could be combined with standard therapies. Thus, the research that is proposed will not only increase the investigators understanding of the impact of negative energy balance on tumor biology, but could change the standard of care and offer a more conservative treatment option for the 50,000 American women who are diagnosed with DCIS each year, as well as a novel adjunct therapy for women with early stage invasive disease.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with intermediate-to-high nuclear grade DCIS or stage I or II breast cancer who elect surgery and who have >3-week lag-time between the start of the intervention and their scheduled surgery;
* Overweight or obese (BMI:25-60);
* English speaking/reading
* Willing to be assigned to either study arm

Exclusion Criteria:

* Have a pre-existing medical condition(s) that preclude adherence to unsupervised exercise;
* Have a current medical condition that affects weight status;
* Has an active malignancy, other than DCIS, invasive breast cancer, or non-melanoma skin cancer;
* Currently enrolled in a weight loss program
* Have received or scheduled to receive neoadjuvant chemotherapy prior to mastectomy or lumpectomy

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-07; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Tumor proliferation | Baseline to Time of Surgery
  Ki-67 will be used to determine tumor proliferation. Ki-67 is a cancer antigen that is found in growing, dividing cells but is absent in the resting phase of cell growth. This characteristic makes Ki-67 a good tumor marker. This test is done on a sample of tumor tissue, to help predict prognosis. High levels of Ki-67 indicate an aggressive tumor and predict a poor prognosis. High scores mean that the cancer cells are growing and dividing at a rapid pace. The Ki-67 scores will be compared between arms.
Weight | Baseline to Time of Surgery
Feasibility | Baseline to Time of Surgery
  Enroll 40 subjects within 2-year study, retain >80% of the sample and completion >70% of contact sessions.

SECONDARY OUTCOMES:
Body Composition | Baseline to Time of Surgery
  Via Dual Energy Absorptiometry (DXA)
Waist Circumference | Baseline to Time of Surgery
Tumor markers | Baseline to Time of Surgery
  Tumor Markers on the CHIEF (Convergence of Hormonal, Inflammatory and Energy-related Factors) Pathway, e.g., Insulin Receptor, Vascular Endothelial Growth Factor (VEGF), Tumor Necrosis Factor alpha (TNF-alpha), Nuclear Factor Kappa Beta (NFKB), caspase-3, as well as various phosphoproteins.
Serum Biomarkers | Baseline to Time of Surgery
  Insulin, leptin, Sex Hormone Binding Globulin, VEGF, TNF-alpha
Gene expression | Baseline to Time of Surgery
  Select genes on the CHIEF pathway as well as ~47,231 curated and putative genes and expressed sequence tags (ESTs)
Dietary Intake | Baseline to Time of Surgery
  24-hour recalls to assess kcal intake as well as intake of fat, protein, and carbohydrate and diet quality
Physical Activity | Baseline to Time of Surgery
  Assessed via accelerometry as well as via questionnaire
Quality of Life | Baseline to Time of Surgery
  Using the FACT-B
Cardiorespiratory Fitness | Baseline to Time of Surgery
  Sub-maximal testing and a modified version of the Naughton Protocol

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Demark-Wahnefried, PhD, RD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Smith KS, Fruge AD, van der Pol W, Caston NE, Morrow CD, Demark-Wahnefried W, Carson TL. Gut microbial differences in breast and prostate cancer cases from two randomised controlled trials compared to matched cancer-free controls. Benef Microbes. 2021 Jun 15;12(3):239-248. doi: 10.3920/BM2020.0098. Epub 2021 Apr 1. PMID 33789551
- [Derived] Fruge AD, Van der Pol W, Rogers LQ, Morrow CD, Tsuruta Y, Demark-Wahnefried W. Fecal Akkermansia muciniphila Is Associated with Body Composition and Microbiota Diversity in Overweight and Obese Women with Breast Cancer Participating in a Presurgical Weight Loss Trial. J Acad Nutr Diet. 2020 Apr;120(4):650-659. doi: 10.1016/j.jand.2018.08.164. Epub 2018 Nov 9. PMID 30420171
- [Derived] Tsuruta Y, Rogers LQ, Krontiras H, Grizzle WE, Fruge AD, Oster RA, Umphrey HR, Jones LW, Azrad M, Demark-Wahnefried W. Exploring effects of presurgical weight loss among women with stage 0-II breast cancer: protocol for a randomised controlled feasibility trial. BMJ Open. 2016 Sep 15;6(9):e012320. doi: 10.1136/bmjopen-2016-012320. PMID 27633639